CLINICAL TRIAL: NCT06365008
Title: Sintilimab Plus FOLFIRI as Salvage Therapy for Patients With Advanced Gastric Cancer: a Prospective Single-arm Phase II Study
Brief Title: Sintilimab Plus FOLFIRI as Salvage Therapy for Patients With Advanced Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYSKY-2024-210-01
Record Dates: First submitted 2024-04-10; First posted 2024-04-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Unresectable/Metastatic Gastric Cancer
Keywords: Sintilimab; FOLFIRI; salvage therapy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients will receive sintilimab 3mg/kg for patients with body weight<60kg or 200mg for patients with body weight ≥ 60kg, plus irinotecan 180mg/m2 intravenous infusion, leucovorin folinate 400mg/m2 intravenous infusion and fluorouracil 400mg/m2 intravenous injection followed by 2400mg/m2 intravenous infusion for 48 hours, repeated every two weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sintilimab+irinotecan+leucovorin folinate+fluorouracil (Experimental): sintilimab 3mg/kg for patients with body weight<60kg or 200mg for patients with body weight ≥ 60kg, plus irinotecan 180mg/m2 intravenous infusion, leucovorin folinate 400mg/m2 intravenous infusion and fluorouracil 400mg/m2 intravenous injection followed by 2400mg/m2 intravenous infusion for 48 hours, repeated every two weeks.
  Interventions: Drug: Sintilimab+irinotecan+leucovorin folinate+fluorouracil

INTERVENTIONS:
Drug: Sintilimab+irinotecan+leucovorin folinate+fluorouracil — sintilimab 3mg/kg for patients with body weight<60kg or 200mg for patients with body weight ≥ 60kg, plus irinotecan 180mg/m2 intravenous infusion, leucovorin folinate 400mg/m2 intravenous infusion and fluorouracil 400mg/m2 intravenous injection followed by 2400mg/m2 intravenous infusion for 48 hours, repeated every two weeks.

SUMMARY:
The combination of immune checkpoint inhibitors and platinum containing dual drugs are more used as a first-line therapeutic approach for patients diagnosed with advanced gastric cancer for its superior efficacy. However, there are no standard recommendations for subsequent treatment after progression on first-line therapy. Here, the investigators conduct this open-label, monocenter, single arm phase II study to evaluate whether sintilimab in combination with irinotecan, leucovorin folinate and fluorouracil can be the salvage therapy for patients diagnosed with unresectable or metastatic gastric cancer progression on first-line therapy. Patients participated in this study will receive sintilimab 3mg/kg for patients with body weight<60kg or 200mg for patients with body weight ≥ 60kg, plus irinotecan 180mg/m2 intravenous infusion, leucovorin folinate 400mg/m2 intravenous infusion and fluorouracil 400mg/m2 intravenous injection followed by 2400mg/m2 intravenous infusion for 48 hours, repeated every two weeks. The primary endpoint is progression-free survival (PFS). The investigators estimated that 40 patients were necessary. Secondary endpoints include overall survival, objective response rate, disease control rate and safety for unresectable or metastatic gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic or locally advanced, unresectable gastric adenocarcinoma confirmed by histology or cytology
2. Progression or toxicity intolerance of first-line treatment
3. Age 18-75 years old
4. ECOG score 0-2
5. Estimated life expectancy of at least 12 weeks
6. Adequate organ and bone marrow function, as follows: Hemoglobin ≥8g/dl, neutrophil absolute count ≥1000/μL, platelets ≥ 75,000 /μL,Total bilirubin ≤1.5 x upper limit of normal (ULN), alkaline phosphatase, aspartate aminotransferase (AST (SGOT) and alanine aminotransferase (ALT (SGPT)) ≤2.5 x ULN (if liver metastasis is present, ≤5 x ULN), Serum albumin≥2.8g/dl, Serum creatinine ≤1.5 x ULN or calculated creatinine clearance >50mL/min (calculated according to Cockcroft Gault formula)
7. International Normalized Ratio (INR) or activated partial thromboplastin time (APTT) <1.5 x ULN (thromboembolic event must be ruled out if D-dimer is abnormal)
8. Negative pregnancy test not more than 7 days before enrollment,Pregnancy tests can only be omitted in women who do not have any reproductive potential (e.g., postmenopausal women, i.e. amenorrhea ≥2 years or prior hysterectomy or bilateral oophorectomy). Fertile women and men must consent to the use of appropriate contraception at the time of enrollment and during study participation for at least 3 months after the last treatment
9. Have sufficient understanding ability and be willing to sign written informed consent

Exclusion Criteria:

1. Pregnant and lactating women
2. The patient has experienced hyperprogression and immunotherapy related grade 3 or above adverse reactions during previous immunotherapy
3. Received antitumor chemotherapy or biotherapy within 28 days prior to the first use of the investigational drug, the total area of previous bone marrow radiation therapy exceeds 30%; the exception is that if it is not the target lesion, palliative radiotherapy is allowed, and the radiotherapy area must be less than 25% of the bone marrow area
4. Suffering from other malignant tumors within the past 5 years or simultaneously
5. Suffering from severe neurological and psychiatric disorders
6. Patients with uncontrolled or symptomatic brain metastases
7. Patients with active autoimmune diseases
8. Immunosuppressive or systemic hormone therapy for immunosuppressive purposes (dose >10mg/ day prednisone or other therapeutic hormone) within 14 days prior to initiation of study therapy
9. Allergies to investigational drugs or excipients
10. Hypertension that cannot be controlled by antihypertensive drugs, coronary heart disease, heart failure, and arrhythmia (QTcF prolongation,>450ms in males and>470ms in females)
11. Severe infection in the 4 weeks prior to initiation of study treatment, including but not limited to hospitalization for complications of infection, bacteremia, or severe pneumoniaOral or intravenous administration of therapeutic antibiotics within 2 weeks prior to initiation of study treatment (patients receiving prophylactic antibiotics, for example, to prevent urinary tract infections or exacerbation of chronic obstructive pulmonary disease are eligible for study participation)
12. Patients with congenital or acquired immune deficiency (such as HIV infection)
13. Have received live attenuated vaccines within 28 days prior to initiation of study treatment, or are expected to require such vaccines during sintilimab treatment or within 60 days after the last administration of sintilimab

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-08 (Estimated); Primary Completion 2027-04-08 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | Undergo imaging examination to evaluate efficacy every 8 weeks ±7 days
  PFS is defined as the time from study enrollment to first disease progression or death, whichever occurs first

SECONDARY OUTCOMES:
Overall survival | From the date of enrollment to the date of death from any cause
  OS is defined as the time from study enrollment to the date of death due to any cause
Objective response rate | Undergo imaging examination to evaluate efficacy every 8 weeks ±7 days
  ORR is defined as the percentage of patients relative to the total of enrolled subjects who achieve a complete response (CR) or partial response (PR) based on CT or MRI scan images
Disease control rate | Undergo imaging examination to evaluate efficacy every 8 weeks ±7 days
  DCR is defined as the percentage of patients relative to the total of enrolled subjects who achieve a complete response (CR) , partial response (PR) or stable disease (SD) based on CT or MRI scan images
Adverse Events | from the date of the first medicine to 28±7 days after the last medicine
  Assessment of Safety and tolerance for sintilimab plus FOLFIRI as salvage therapy in patients with unresectable/metastatic gastric cancer, including incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI CTC AE Version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Qiong Yang, Doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University; Yajing Liu, Doctor, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital,Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No